CLINICAL TRIAL: NCT02961153
Title: Epidemiology of Death in the PICU of Southeast China
Brief Title: Mortality in Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Guoping Lu, Director of pediatric Emergency and Critical Care Center. Children's Hospital Fudan University;Director of AHA Training Center for pediatric life support. Children's Hospital Fudan University, Children's Hospital of Fudan University
Other Study IDs: fdpicu-01
Record Dates: First submitted 2016-10-26; First posted 2016-11-10 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Intensive Care Units, Pediatric
MeSH Terms: interventions — Death Domain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: death

SUMMARY:
With the development of national economy and medical technology, patients can extend life rely on high-end medical facilities. At the same time, the continued treatment cannot bring benefits to children, even resulting in poor quality of life of children and bringing high medical costs. This makes the limited medical resources are unreasonable distributed. Research showed that PICU mortality rate halved over ten years ago, but the data did not include death cases who left hospital before death. However, the death number of out-hospital were more than death in-hospital. Therefore, the data cannot actually reflect China's mortality rate of PICU. The reason analysis was limited to the cause of the disease, and does not take the social, economic factors into account. This study include eight PICUs of children's Hospital PICU. Critically ill patients are prospectively studied from death risk factors, admission status, disease diagnosis, severity of illness, analyzing of the risk factors of death from disease diagnosis and death risk factors. In addition, we will illuminate the relationship of death and economic factor, especially for who died out-hospital after withdraw or stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* ALL patients admitted to the PICU of eight study centers

Exclusion Criteria:

* Postoperative monitoring of patients with stable hemodynamics
* PCIS score >90 and not up to the United States PICU admission standards

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ALL patients admitted to the PICU of eight study centers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Pediatric Critical Illness Score（PCIS） | first 24 hours after admission
Pediatric Risk of Mortality score (PRISM III) | 24 hours
Pediatric logistic organ dysfunction (PELOD) score | 24hour

SECONDARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: LU guoping, doctor, Principal Investigator — Children's Hhospital of Fudan University
Locations (1):
- Children'S Hosptial of Fuan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No